CLINICAL TRIAL: NCT07168213
Title: Comparison of Two SpO2 Targets With Two Different Oximeters - Impact on FiO2 During Nasal High Flow Oxygen Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2026-4432
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Oxygen Delivery; Acute Respiratory Failure; High Flow Oxygen Therapy; Hypoxemic Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nonin oximeter with a 90% SpO2 target (Experimental): During this periods , oxygen through high flow nasal therapy a will be administered in an manual titration to reach 90% of SpO2.
  Interventions: Device: Manual FiO2 titration with Nonin oximeter (SpO2 target 90%)
- Philips oximeter with a 90% SpO2 target (Experimental): During this periods , oxygen through high flow nasal therapy a will be administered in an manual titration to reach 90% of SpO2.
  Interventions: Device: Manual FiO2 titration with Philips oximeter (SpO2 target 90%)
- Nonin oximeter with a 94% SpO2 target (Experimental): During this periods , oxygen through high flow nasal therapy a will be administered in an manual titration to reach 94% of SpO2.
  Interventions: Device: Manual FiO2 titration with Nonin oximeter (SpO2 target 94%)
- Philips oximeter with a 94% SpO2 target (Experimental): During this periods , oxygen through high flow nasal therapy a will be administered in an manual titration to reach 94% of SpO2.
  Interventions: Device: Manual FiO2 titration with Philips oximeter (SpO2 target 94%)

INTERVENTIONS:
Device: Manual FiO2 titration with Philips oximeter (SpO2 target 90%) — FiO2 titration to reach the SpO2 target (set at 90%) with Philips oximeter
  Arms: Philips oximeter with a 90% SpO2 target
Device: Manual FiO2 titration with Nonin oximeter (SpO2 target 90%) — FiO2 titration to reach the SpO2 target (set at 90%) with Nonin oximeter
  Arms: Nonin oximeter with a 90% SpO2 target
Device: Manual FiO2 titration with Philips oximeter (SpO2 target 94%) — FiO2 titration to reach the SpO2 target (set at 94%) with Philips oximeter
  Arms: Philips oximeter with a 94% SpO2 target
Device: Manual FiO2 titration with Nonin oximeter (SpO2 target 94%) — FiO2 titration to reach the SpO2 target (set at 94%) with Nonin oximeter
  Arms: Nonin oximeter with a 94% SpO2 target

SUMMARY:
Several factors can influence oxygenation monitoring and respiratory support through oxygen therapy: the type of oximeter used, skin pigmentation, and the oxygenation target. It is essential to have an accurate measurement of SpO2 in order to optimize the flow of oxygen or FiO2 administered to patients. The question arises as to the impact of these confounding factors on the FiO2 set during high-flow nasal oxygen therapy. The aim of the study is to evaluate the impact of the oxygenation target and the oximeter used on FiO2 in patients receiving high-flow nasal oxygen therapy.

DETAILED DESCRIPTION:
The oximeters evaluated will be the Nonin (Plymouth, MN) and the Philips (Eindhoven, Netherlands). Two SpO2 targets will be evaluated: 90% and 94%.

A total of four 10-minute periods will be performed in randomized order: Nonin 90, Nonin 94, Philips 90, and Philips 94.

At the end of each 10-minute period, arterial gas will be collected through the arterial catheter.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Admiitted in intensive care unit
* Presence of an arterial catheter
* Ongoing on high flow nasal oxygen therapy with SpO2 between 88 and 100% with a FiO2 between 40 and 80% with the usual oximeter .

Exclusion Criteria:

* No SpO2 signal with oximeter in use
* False nails or nail polish
* Methemoglobinemia >0.015 on last available arterial gas
* Patient in isolation (multi-resistant bacteria, C-Difficile, SARS-CoV-2 ...)
* Expected to use another respiratory support within two hour of inclusion (NIV or mechanical ventilation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
FiO2 | Mean FiO2 in the two last minute of each study period between minute 8 and 10
  FiO2 at the end of each study period (last minute average) to reach SpO2 target to reach SpO2 target with specific oximeter

SECONDARY OUTCOMES:
Difference between SpO2 and SaO2 | assessed up to 10 minutes - at the same of the arterial blood gases punction
  Difference (%) between SpO2 from each oximeter and SaO2 (% of SaO2 overestimation and underestimation for each oximeter)
High flow weaning criteria | Mean FiO2in the two last minute of each study period (between minute 8 and 10)
  Percentage of patient whose average FiO2 level below 40%
Intensive care unit transfert criteria | Mean FiO2in the two last minute of each study period (between minute 8 and 10)
  Percentage of patients whose average FiO2 level over 60%
Intubation criteria | Mean FiO2in the two last minute of each study period (between minute 8 and 10)
  Percentage of patients whose average FiO2 level over 80%
Mean difference on oxymeter | assessed up to 10 minutes - at the same of the arterial blood gases punction
  Mean (±SD) of the gaps between the different oximeters tested

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No